CLINICAL TRIAL: NCT01012089
Title: Study of the Pharmacokinetics of Daptomycin in Children With Renal Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Collaborators: Cubist Pharmaceuticals LLC, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2375
Record Dates: First submitted 2009-11-09; First posted 2009-11-11 (Estimated); Results first posted 2018-06-06 (Actual); Last update posted 2018-06-06 (Actual); Status verified 2018-05

CONDITIONS: Chronic Kidney Disease; Bacterial Infection
Keywords: Hemodialysis; Peritoneal dialysis; Daptomycin; Pharmacokinetics
MeSH Terms: conditions — Renal Insufficiency, Chronic; Bacterial Infections | interventions — Daptomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Daptomycin (Experimental): Pediatric patients on hemodialysis or peritoneal dialysis with suspected or confirmed infection and who were receiving standard of care antibiotics were also eligible to receive a single dose of daptomycin 5mg/kg IV. Serial blood draws were obtained to assess daptomycin pharmacokinetics
  Interventions: Drug: Daptomycin

INTERVENTIONS:
Drug: Daptomycin — Daptomycin IV 5 mg/kg one time dose
  Other Names: Cubicin

SUMMARY:
The purpose of this study is to:

1. Study the pharmacokinetics and safety of daptomycin in children on hemodialysis (HD) and peritoneal dialysis (PD).
2. Determine urine, HD and PD clearance of daptomycin.

DETAILED DESCRIPTION:
Infectious and sepsis events are one of the most common complications in children with chronic kidney disease. The incidence is highest in children with an access for dialysis, especially in those with catheters. Staphylococcal species account for more than 50% of access infections (ranging from 58-77%). Failure to clear the infection results in loss of dialysis access.

Daptomycin is a new antibiotic that provides coverage against most gram positive bacteria including methicillin-resistant staphylococci, vancomycin-intermediate Staphylococcus aureus, and vancomycin-resistant enterococci. The pharmacokinetics of daptomycin in children on dialysis, a group of patients who may need the medication the most, remains unknown.

Children on HD or PD with suspected or confirmed infections due to gram-positive bacteria and who are concurrently treated with standard of care antibiotics will be considered for this study. Each patient will be given a onetime dose of Cubicin (daptomycin). After receiving daptomycin, serial blood samples along with dialysis effluent and urine (obtained from non-anuric patients) will be collected to evaluate the pharmacokinetic profile of the drug.

ELIGIBILITY:
Inclusion Criteria:

* Children who are between 12-17 years of age who are either on HD or PD and whom the Pediatric Nephrology Section of the OU Children's Physicians Clinics provide care.
* In addition to children on chronic HD and PD therapy, patients newly initiated on HD and PD will also be recruited for this study.
* Patients with suspected or confirmed cases of dialysis related infection from gram-positive bacteria and who are receiving standard of care antibiotics.
* Patients will be eligible for enrollment if they were admitted as an inpatient to the Children's hospital or as an outpatient to the dialysis clinic

Exclusion Criteria:

* Patients > 17 years of age
* Patients < 12 years of age
* Total amount of blood drawn as part of standard of care and for pharmacokinetic analysis exceeds 3 ml/kg over an 8 week period
* Taking an HMG CoA reductase inhibitor within 7 days of daptomycin administration
* Having used daptomycin in the 30 days preceding study entry
* Participating in any experimental procedure in the 30 days preceding study
* A history of muscular disease or neurological disease
* Baseline creatine phosphokinase (CPK) values equal to or greater than 1.5 times the upper limit of normal (normal range 65-370 IU/L)
* Hemoglobin < 9 g/dl
* Hemodynamic instability within 72 hours before study enrollment
* Female subjects with a positive pregnancy test or failure to take a pregnancy test

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 6 (Actual)
Dates: Start 2009-11; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Teresa V Lewis, Pharm.D., Principal Investigator — University of Oklahoma; Martin A Turman, M.D., Ph.D., Principal Investigator — University of Oklahoma
Locations (1):
- The Children's Hospital at the University of Oklahoma Medical Center, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Daptomycin
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Daptomycin Hemodialysis: Daptomycin: Daptomycin IV 5 mg/kg one time dose to patient receiving intermittent hemodialysis on MWF
- Daptomycin Peritoneal Dialysis: Daptomycin: Daptomycin IV 5 mg/kg one time dose to patient receiving continuous cycling peritoneal dialysis
- Total: Total of all reporting groups
Arm/Group | Daptomycin Hemodialysis | Daptomycin Peritoneal Dialysis | Total
Number analyzed (Participants) | 3 | 3 | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3 | 3 | 6
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 15.3 [14 to 17] | 13.7 [12 to 15] | 14.5 [12 to 17]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 3 | 2 | 5
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Maximum Plasma Concentration (Cmax)
Time Frame: 0, 0.5, 2, 3, 4.5 6, 24, and 48 hours post dose
Population: The PK analysis population were pediatric dialysis patients who had either confirmed or suspected infection who received appropriate antibiotic treatment of their infection along with a single dose of daptomycin
Measure: Mean (Full Range); unit: mg/L
Groups:
- Daptomycin Hemodialysis: Pediatric hemodialysis patients who received a one time dose of Daptomycin IV 5 mg/kg administered prior to a hemodialysis session
- Daptomycin Peritoneal Dialysis: Pediatric peritoneal patients who received a one time dose of Daptomycin IV 5 mg/kg administered prior to a peritoneal dialysis session
Arm/Group | Daptomycin Hemodialysis | Daptomycin Peritoneal Dialysis
Number analyzed (Participants) | 3 | 3
mg/L | 42.4 [36.1 to 46.5] | 66.5 [45.1 to 97.8]

2. Primary Outcome: Area Under the Concentration Time Curve From Time Zero to 24 Hours (AUC0-24)
Time Frame: 0, 0.5, 2, 3, 4.5, 6, and 24 hours post dose
Population: as for outcome 1
Measure: Mean (Full Range); unit: mg∙hr/L
Arm/Group | Daptomycin Hemodialysis | Daptomycin Peritoneal Dialysis
Number analyzed (Participants) | 3 | 3
mg∙hr/L | 388 [323 to 429] | 708 [525 to 944]

3. Primary Outcome: Area Under the Concentration Time Curve From Time Zero to 48 Hours (AUC0-48)
Time Frame: 0, 0.5, 2, 3, 4.5 6, 24, and 48 hours post dose
Population: as for outcome 1
Measure: Mean (Full Range); unit: mg∙hr/L
Arm/Group | Daptomycin Hemodialysis | Daptomycin Peritoneal Dialysis
Number analyzed (Participants) | 3 | 3
mg∙hr/L | 557 [454 to 617] | 1051 [804 to 1412]

4. Primary Outcome: Area Under the Concentration Time Curve From Time Zero to Infinity (AUC0-∞)
Time Frame: 0, 0.5, 2, 3, 4.5, 6, 24, and 48 hours post dose
Population: as for outcome 1
Measure: Mean (Full Range); unit: mg∙hr/L
Arm/Group | Daptomycin Hemodialysis | Daptomycin Peritoneal Dialysis
Number analyzed (Participants) | 3 | 3
mg∙hr/L | 734 [579 to 874] | 1477 [1142 to 2127]

5. Primary Outcome: Volume of Distribution at Steady State (Vss)
Description: The theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired blood concentration of a drug
Time Frame: 0, 0.5, 2, 3, 4.5, 6, 24, and 48 hours post dose
Population: as for outcome 1
Measure: Mean (Full Range); unit: L
Arm/Group | Daptomycin Hemodialysis | Daptomycin Peritoneal Dialysis
Number analyzed (Participants) | 3 | 3
L | 5.89 [4.68 to 6.99] | 6.38 [6.23 to 6.49]

6. Primary Outcome: Elimination Rate Constant (Ke)
Time Frame: 0, 0.5, 2, 3, 4.5, 6, 24, and 48 hours post dose
Population: as for outcome 1
Measure: Mean (Full Range); unit: hr-1
Arm/Group | Daptomycin Hemodialysis | Daptomycin Peritoneal Dialysis
Number analyzed (Participants) | 3 | 3
hr-1 | 0.0053 [0.00358 to 0.00777] | 0.00848 [0.00848 to 0.00848]

7. Primary Outcome: Total Drug Clearance (CLtotal)
Description: The rate at which a drug substance is removed from the body
Time Frame: 0, 0.5, 2, 3, 4.5, 6, 24, and 48 hours post dose
Population: as for outcome 1
Measure: Mean (Full Range); unit: mL/hr
Arm/Group | Daptomycin Hemodialysis | Daptomycin Peritoneal Dialysis
Number analyzed (Participants) | 3 | 3
mL/hr | 177 [150 to 221] | 170 [143 to 208]

8. Primary Outcome: Drug Clearance Due to Dialysis (CLdialysis)
Description: The rate at which a drug substance is removed from the body due to dialysis therapy
Time Frame: 0, 0.5, 2, 3, 4.5, 6, 24, and 48 hours post dose
Population: as for outcome 1
Measure: Mean (Full Range); unit: mL/hr
Arm/Group | Daptomycin Hemodialysis | Daptomycin Peritoneal Dialysis
Number analyzed (Participants) | 3 | 3
mL/hr | 670 [646 to 690] | 21 [18 to 23]

ADVERSE EVENTS:
Time Frame: Safety assessments were performed on study "Day 0", "Day 1", "Day 2". Serum CPK and standard clinical laboratory evaluations were obtained at baseline and at the end of study "Day 0". A telephone follow-up was also conducted by study personnel at Day 7, 14, 21 and 28 post study drug administration to continue follow-up of potential adverse events.
Groups:
- Daptomycin Peritoneal Dialysis: Pediatric dialysis patients who received a one time dose of Daptomycin: Daptomycin IV 5 mg/kg administered prior to a peritoneal dialysis session
Arm/Group | Daptomycin Peritoneal Dialysis | Daptomycin Hemodialysis
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 0/3 | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No